CLINICAL TRIAL: NCT04558827
Title: Feasibility Study of a Low-Carb/Time-restricted Feeding Protocol in Insulin-Using Type 2 Diabetics
Brief Title: Low-Carb/Time-restricted Feeding Protocol in Insulin-Using Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0140; A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 4/20/2020 (Other: UW Madison)
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes
Keywords: low carbohydrate diet; time restricted feeding; insulin sensitivity
MeSH Terms: conditions — Intermittent Fasting; Insulin Resistance | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Carb / Time Restricted Feeding (Experimental): Participants will eat a low carbohydrate diet (30-60 grams) in a time restricted feeding window (2 meals within 8 hours) daily for the duration of the study (6 months).
  Interventions: Other: Low Carbohydrate Diet; Other: Time Restricted Feeding

INTERVENTIONS:
Other: Low Carbohydrate Diet — Dietary choices are counseled to come primarily from lean meats, eggs, nuts, seeds, vegetables and berries.
Other: Time Restricted Feeding — Participants will be asked to have 2 meals within an 8 hour period, preferably before 2pm.
  Other Names: Intermittent Fasting

SUMMARY:
The current paradigm of Type 2 Diabetes treatment relies heavily on expensive pharmacotherapy even though lifestyle factors are at the root of the condition. This study is designed to assess the feasibility of a low carbohydrate diet coupled with a time restricted feeding intervention to improve participant sensitivity, reducing their need for insulin. 20 participants will be invited to enroll from the 20 S Park St Clinic in Madison, WI and remain on study for up to 6 months.

DETAILED DESCRIPTION:
The investigators will perform a prospective cohort study of 20 insulin-using Type 2 diabetics who have primary care providers at 20 S Park St Clinic. Participants will be recruited from the Internal Medicine practices at the clinic. The subjects will meet with Dr. Zimmermann (Study Clinician) to review time restricted feeding and low-carbohydrate diets as well as a strategy for decreasing insulin doses. Calls from Dr. Zimmermann's clinic nurse will occur daily until blood glucose levels stabilize to manage insulin decrease.

Participants will complete monthly logs of food intake times and meet with a dietician twice during the 6-month study. Diabetes medication use will be reviewed, and hemoglobin A1c will be measured, at baseline and at 3 and 6 months. The participants' non-diabetic medical care will continue to be managed through their primary care physicians (PCPs).

Specific Aims:

* Demonstrate feasibility of the low carbohydrate/time restricted feeding (LC/TRF) protocol

  * Feasibility will be assessed based on participant compliance with time-restricted feeding and recommended carbohydrate intake, clinician time and clinic resources
* Determine effectiveness of the LC/TRF protocol on diabetes care and quality of life

  * Effectiveness on diabetes care will be evaluated using changes in A1c, insulin use, BMI, patient quality of life, and adverse events including hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient of a primary care provider at 20 S Park Internal Medicine Clinic
* Insulin using type 2 diabetic
* Using glargine or detemir insulin for basal insulin dosing
* Self-administering insulin
* Hemoglobin A1c 7-10%.
* Stable diabetes regimen for >3 months
* Demonstrated reliability with glucose monitoring, A1c checks
* BMI 25-35

Exclusion Criteria:

* History consistent with type 1 diabetes
* Using concentrated insulin (U200 or U300)
* Living in a skilled nursing facility
* Unwilling or unable to do frequent (3x daily) blood glucose checks
* eGFR (estimated glomerular filtration rate) < 30 mL/min per 1.73 m2
* Currently on steroids or warfarin
* Hospitalized within 3 months
* Symptomatic heart failure
* Weight Loss >10% in last six months
* History of organ transplantation
* Pregnant/trying to become pregnant/breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Intervention: Changes in Hemoglobin A1c | baseline, 3 months, 6 months
  Changes in A1c will be measured at baseline, 3 and 6 month MD visits. Data will be extracted from HealthLink by chart review. Comparisons will be made between post-intervention A1c scores and baseline scores, at 1 month and at 3 months using paired t-tests to detect whether patients experienced a positive outcome.
Effectiveness of Intervention: Changes in Insulin Dosage | baseline, 3 months, 6 months
  Changes in insulin dosage will be measured at baseline, 3 and 6 month MD visits. Data will be extracted from HealthLink by chart review.

SECONDARY OUTCOMES:
Participant Satisfaction | 3 months, 6 months
  Participant satisfaction with the protocol will be assessed at 3 and 6 months. This will include questions about difficulty, barriers to implementation, and impact on family. Quantitative and qualitative analysis will be performed to determine barriers and facilitators to maintaining TRF and low carbohydrate diet. Semi-structured phone interviews will be performed with 10 of the patients (5 who maintained the LC/TRF protocol and 5 who did not) to understand the impact of the TRF and low carbohydrate diet on their daily lives and determine barriers and facilitators. Interviews will be transcribed and thematic analysis will be performed.
Change in Appraisal of Diabetes Scale (ADS) Score | baseline, 3 months, 6 months
  Participant quality of life (QoL) will be assessed at baseline, 3 and 6 months with the Appraisal of Diabetes Scale (ADS). The ADS is a validated tool to measure patients' appraisal of how well they can care for their diabetes and its impact on their life. It is a 7-item survey with each question scored on a likert scale (1-5) for a total range of possible scores 7-35, where lower scores indicate better QoL. Statistical analysis will be performed using paired t-tests or non-parametric methods based on distribution to evaluate ADS changes over time.
Clinic-level feasibility: Average Hours of Support Time per Participant | up to 6 months
  MD and RD clinic time along with RN phone support will be logged with each encounter to provide a quantitative assessment of the resources required to implement this type of intervention on a clinic scale. Descriptive statistics with means and standard deviations per patient will be calculated for each class of health care provider.
Effectiveness of Intervention: Changes in BMI | baseline, 3 months, 6 months
  Changes in BMI will be measured at baseline, 3 and 6 month MD visits. Data will be extracted from HealthLink by chart review. Weight and height will be combined to report BMI in kg/m^2.
Feasibility: Percent of days where food was eaten within the target timeframe | up to 6 months
  Participant compliance with time-restricted feeding will be evaluated using monthly journals logging first and last food intake each day. The journals will be mailed to Dr. Zimmermann via pre-addressed/stamped security envelopes or brought to appointments. Time-restricted feeding compliance will be calculated using descriptive statistics to determine the % of days where all food was eaten within the target timeframe. Analysis will be done for all data available, data from participants with logs for >50% of days, and participants with logs for >75% of days.
Feasibility: Average Daily Calories | up to 6 months
  Participant compliance with recommended carbohydrate intake will be evaluated based on data from the registered dietitian (RD) dietary review. RD will calculate daily grams of carbohydrate and total calories. Compliance will be calculated with descriptive statistics for % of days compliant with <30g, 30-60g, >60g of carbohydrates as well as average daily calories.
Feasibility: Percent of day compliant with Carbohydrate target | up to 6 months
  Participant compliance with recommended carbohydrate intake will be evaluated based on data from the registered dietitian (RD) dietary review. RD will calculate daily grams of carbohydrate and total calories. Compliance will be calculated with descriptive statistics for % of days compliant with <30g, 30-60g, >60g of carbohydrates as well as average daily calories.

CONTACTS AND LOCATIONS:
Overall Officials: David Feldstein, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (3):
- United States (3):
  - UW Health Union Corners Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - UW Health West Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No